CLINICAL TRIAL: NCT01387295
Title: Intra-hepatic Chemotherapy With Oxaliplatin Every Second Week in Combination With Systemic Capecitabine in Patient With Non-resectable Liver Metastases From Breast Cancer A Phase II Trial in Patients With Limited Extrahepatic Disease
Brief Title: Intra-hepatic Chemotherapy in Patients With Liver Metastases From Breast Cancer and Limited Extrahepatic Disease
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Dorte Nielsen (Other)
Responsible Party: Sponsor-Investigator, Dorte Nielsen, Responsible Party was entered in the old format as Dorte Nielsen, professor DMSci, Department of Oncology, Herlev Hospital., Herlev Hospital
Organization: Herlev Hospital (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MA 0918
Record Dates: First submitted 2011-05-31; First posted 2011-07-04 (Estimated); Results first posted 2023-12-11 (Actual); Last update posted 2023-12-11 (Actual); Status verified 2023-03

CONDITIONS: Metastatic Breast Cancer; Liver Metastases
Keywords: breast cancer; liver metastases; intrahepatic chemotherapy
MeSH Terms: conditions — Breast Neoplasms | interventions — Oxaliplatin; Capecitabine; Trastuzumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- chemotherapy (Experimental)
  Interventions: Drug: oxaliplatin, capecitabine, trastuzumab

INTERVENTIONS:
Drug: oxaliplatin, capecitabine, trastuzumab — Oxaliplatin intrahepatic capecitabine and trastuzumab systemic
  Other Names: HAI

SUMMARY:
This is a phase II trial evaluating intra-hepatic chemotherapy with oxaliplatin every second week in combination with systemic capecitabine and in patients with a HER2-positive tumour in combination with trastuzumab (Herceptin®) in patient with non-resectable liver metastases from breast cancer.

Only patients with limited extrahepatic disease are included.

ELIGIBILITY:
Inclusion Criteria:• Informed consent

* Age > 18 years
* Performance status 0-1; expected survival ≥ 3 months
* Patient with histologically or cytologically confirmed locally advanced or metastatic adenocarcinoma of the breast
* Liver metastases not suitable for local treatment
* Extrahepatic disease should be determined by PET-CT-scan.
* No progression on treatment with capecitabine.
* Prior treatment with taxane (adjuvant or for metastatic disease)
* Metastases < 70 % of the liver
* Neutrophile granulocytes > 1.5 x 109/l og thrombocytes > 100 x 109/l
* Bilirubin < 2.0 x UNL (upper normal limit).
* Creatinine-clearance > 30 ml/min.
* INR < 1.6.
* If the patient is HER2-positive:Baseline LVEF ≥ 50 %

Exclusion Criteria:

* History of chemotherapy within the 4-week period prior to the start of trial medication
* Other current or prior malignant disease except adequately treated and cured carcinoma in situ of the cervix or squamous cell carcinoma of the skin.
* Previous treatment with oxaliplatin
* Cytotoxic or experimental treatment within a 14 days period before start of trial medication
* The patient is not allowed to participate in other clinical trials.
* Any clinical symptoms suggesting peripheral neuropathy < or equal to grade 2 or CNS metastases (In case of clinical suspicion on CNS metastases a MR or CT scan should be performed within 4 weeks before inclusion
* Other severe medical conditions e.g. severe cardial disease or AMI < 1 year
* Presence of diseases which prevent oral therapy.
* Patients with uncontrolled infection
* Pregnant or lactating women
* Women capable of childbearing not using a sufficient non-hormonal method of birth control
* Patients not able to understand the treatment or to collaborate.
* Prior serious or unsuspected reaction after treatment with fluoropyrimidine
* Known prior hypersensitivity reactions to the agents

If the patient is HER2-positive:

* Dyspnoea in due to complication related to malignant disease e.g.lung metastases with lymphangitis or other conditions with need of supportive oxygen.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2010-04; Primary Completion 2017-05-01 (Actual); Study Completion 2017-09-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Dorte Nielsen, Professor, Principal Investigator — professor
Locations (1):
- Herlev Hospital, Herlev, Denmark

REFERENCES:
- [Result] Lindgaard SC, Brinch CM, Jensen BK, Norgaard HH, Hermann KL, Theile S, Larsen FO, Jensen BV, Michelsen H, Nelausen KM, Holm VH, Ekblad L, Soerensen PG, Nielsen DL. Hepatic arterial therapy with oxaliplatin and systemic capecitabine for patients with liver metastases from breast cancer. Breast. 2019 Feb;43:113-119. doi: 10.1016/j.breast.2018.12.002. Epub 2018 Dec 5. PMID 30544058

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Chemotherapy
Started | 38
Completed | 38
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Chemotherapy
Number analyzed (Participants) | 38
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 30
  >=65 years | 8
Age, Continuous [Median (Full Range); unit: years] | 54.5 [31 to 72]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 38
  Male | 0
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  Denmark | 38

OUTCOME MEASURES:

1. Primary Outcome: Response Rate
Description: Number of patients with complete or partial response in the liver (RECIST version 1.1). Only patients with measurable disease are included in the protocol. Response rate number of patients with CR + PR divided with total number.
  Per Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0) for target lesions and assessed by MRI: Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions,
Time Frame: up to 24 months from baseline
Measure: Count of Participants; unit: Participants
Arm/Group | Chemotherapy
Number analyzed (Participants) | 38
Participants
  CR | 2
  PR | 13
  SD | 21
  PD | 1
  NE | 1

2. Secondary Outcome: Number of Patients Suitable for Local Therapy (Radiofrequency)
Description: Total number of patients receiving RF treatment or surgical treatment
Time Frame: upon completion of treatment, an average of 7 months
Measure: Count of Participants; unit: Participants
Arm/Group | Chemotherapy
Number analyzed (Participants) | 38
Participants | 2

3. Secondary Outcome: Survival
Description: All patients in intent-to-treat population , calculated from start of treatment to death of any course
Time Frame: up to 7 years
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Chemotherapy
Number analyzed (Participants) | 38
months | 24.0 [17.2 to 30.8]

4. Secondary Outcome: Adverse Events
Description: Number of participants with at least 1 AE related to study treatment - The details on which AEs occured are listed in the Adverse Event section below
Time Frame: from start of treatment to 28 days after last treatment, an average of 7 months
Population: All patients who received at least one dose of study drug are evaluable for toxicity. CTC version 3.0 will be used.
Measure: Count of Participants; unit: Participants
Arm/Group | Chemotherapy
Number analyzed (Participants) | 38
Participants | 38

5. Secondary Outcome: PFS
Description: From start of therapy to progression or death of any cause.
Time Frame: up to 6 years
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Chemotherapy
Number analyzed (Participants) | 38
months | 12.8 [6.9 to 18.6]

ADVERSE EVENTS:
Time Frame: Adverse Events were collected from informed consent to 28 days after last treatment, an average of 7 months. All-Cause Mortality was assessed through study completion, up to 7 years
Arm/Group | Chemotherapy
All-Cause Mortality (participants affected / at risk) | 33/38
Serious Adverse Events (participants affected / at risk) | 8/38
Other Adverse Events (participants affected / at risk) | 38/38
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Chemotherapy (N=38)
Morphine toxication (Injury, poisoning and procedural complications) | 1 (1)
Pulmonary embolism (Vascular disorders) | 2 (2)
Fever (General disorders) | 1 (1)
gallbladder stone (Hepatobiliary disorders) | 1 (1)
Diabetes mellitus (Metabolism and nutrition disorders) | 1 (1)
Infection (Infections and infestations) | 3 (3)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Chemotherapy (N=38)
Alanine aminotransferase increased (Investigations) | 15 (38)
Aspartate aminotransferase increased (Investigations) | 19 (77)
Alkaline phosphatase increased (Investigations) | 14 (34)
Hyperbilirubinaemia (Investigations) | 3 (8)
Thrombocytopenia (Investigations) | 17 (82)
Neutropenia (Investigations) | 15 (25)
Anaemia (Blood and lymphatic system disorders) | 9 (12)
Dysaesthesia (Nervous system disorders) | 35 (304)
Peripheral motor neuropathy (Nervous system disorders) | 11 (41)
Peripheral sensory neuropathy (Nervous system disorders) | 29 (179)
Allergic reaction (General disorders) | 3 (6)
Fatigue (General disorders) | 30 (159)
Fever (General disorders) | 9 (12)
Pain (General disorders) | 23 (59)
Diarrhoea (Gastrointestinal disorders) | 21 (55)
Stomatitis (Gastrointestinal disorders) | 21 (62)
Nausea (Gastrointestinal disorders) | 34 (119)
Vomiting (Gastrointestinal disorders) | 20 (36)
Dyspepsia (Gastrointestinal disorders) | 5 (12)
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 33 (184)
Alopecia (Skin and subcutaneous tissue disorders) | 6 (6)
Myalgia (Musculoskeletal and connective tissue disorders) | 5 (12)
Arthralgia (Musculoskeletal and connective tissue disorders) | 4 (8)
Anorexia (Metabolism and nutrition disorders) | 24 (91)
infection (Infections and infestations) | 2 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2012-11-08): https://cdn.clinicaltrials.gov/large-docs/95/NCT01387295/Prot_SAP_000.pdf